CLINICAL TRIAL: NCT07051928
Title: A Prospective, Observational, Single Arm, Multi-site, Pilot Study of Atezolizumab in Non-oncogene Addicted Advanced Nsclc Patients With Pd-l1 Tps ≥ 50%, With Longitudinal Assessment of C-FLIP Expression of Monocytic Myeloid-derived Suppressor Cells
Brief Title: Study of Atezolizumab in Advanced Non-oncogene-addicted NSCLC With PD-L1 ≥50%, Including Longitudinal c-FLIP Assessment in Monocytic MDSCs.
Acronym: FLIP-IMMUNO
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7742
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Immunotherapy; Lung cancer; Atezolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: c-FLIP expression on MDSC — Longitudinal c-FLIP expression on circulating MDSC

SUMMARY:
Prospective, observational, multi-site, single arm, exploratory pilot study, designed to prospectively assess the relationship between basal c-FLIP expression in M-MDSCs with clinical outcomes in patients treated with anti-PD-L1 monotherapy in a 1L mNSCLC setting, as well as evaluate changes in c-FLIP during treatment and correlate those changes with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of signing Informed Consent Form
* ECOG Performance Status of 0-2
* Advanced/metastatic NSCLC without prior treatment in the metastatic setting
* Tumor PD-L1 expression with a TPS ≥ 50%, documented through local testing
* Measurable disease per RECIST v1.1
* Adequate hematologic and end-organ function

Exclusion Criteria:

* Ineligibility to receive first line immunotherapy treatment
* Patients with driver mutations amenable to molecular targeted therapies in I-line according to the indications of the AIFA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age ≥ 18 years with ECOG Performance Status of 0 to 2 who have previously untreated metastatic non-oncogene addicted PD-L1-selected NSCLC (TPS ≥50%)
Sampling Method: Non-Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Disease-control Rate (DCR) | 24 months
  Disease-control rate at 12 weeks based on basal c-FLIP expression on MDSC

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  Median Progression-free Survival among subgroups defined according to c-FLIP expression in M-MDSC at baseline
Overall Survival (OS) | 24 months
  Median overall survival among subgroups defined according to c-FLIP expression in M-MDSC at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Bria, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riley JS, Hutchinson R, McArt DG, Crawford N, Holohan C, Paul I, Van Schaeybroeck S, Salto-Tellez M, Johnston PG, Fennell DA, Gately K, O'Byrne K, Cummins R, Kay E, Hamilton P, Stasik I, Longley DB. Prognostic and therapeutic relevance of FLIP and procaspase-8 overexpression in non-small cell lung cancer. Cell Death Dis. 2013 Dec 5;4(12):e951. doi: 10.1038/cddis.2013.481. PMID 24309938